CLINICAL TRIAL: NCT06440811
Title: Efficacy and Safety of Neoadjuvant Nivolumab Plus SOX Versus Nivolumab Plus FLOT in Patients With HER2-negative Gastric and Gastroesophageal Junction Adenocarcinoma: A Multicentre, Open-Label, Prospective Cohort Study
Brief Title: Efficacy and Safety of Neoadjuvant Nivolumab Plus SOX Versus Nivolumab Plus FLOT in Patients With HER2-negative Gastric and Gastroesophageal Junction Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: loong-101
Record Dates: First submitted 2024-04-06; First posted 2024-06-04 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Immune-related Adverse Event; Chemotherapeutic Toxicity; Gastric or Gastroesophageal Junction Adenocarcinoma
Keywords: neoadjuvant chemotherapy; Nivolumab; SOX; FLOT; locally advanced; HER-negative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — Tumor tissues and adjacent tissues were obtained from every patient in these two cohorts. Thess tissues would be used for pathological histologyfor (Hematoxylin and eosin (H&E)) and cluadin18.2 identified by Immunohistochemistry (IHC) and tertiary lymphoid structures (TLS) identified by Immunofluorescence.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FLOT+nivolumab: Patients in the FLOT group received 4 cycles of standard FLOT chemotherapy, the FLOT chemotherapy cycle consists of: day 1: intravenous 5-FU 2600 mg/m² inserted through a peripherally inserted central catheter (PICC) for 24 hours intravenous folic acid 200 mg/m2 intravenous oxaliplatin 85 mg/m² intravenous docetaxel 50 mg/m². The next cycle of chemotherapy was repeated on day 15. Nivolumab (360 mg) was administered intravenously (IV) over 30 minutes once every 3 weeks for 6 weeks (1 cycle, 2 doses).
- SOX+nivolumab: Patients in the SOX group received 3 cycles of S-1 + OXA chemotherapy prior to radical gastrectomy.The SOX chemotherapy cycle consists of: day 1: intravenous OXA 130 mg/m² days 1-14: oral S-1 80 mg/m², 2 times/Day. Repeat next chemotherapy on day 22. Nivolumab (360 mg) was administered intravenously (IV) over 30 minutes once every 3 weeks for 6 weeks (1 cycle, 2 doses).

SUMMARY:
The goal of the study is to learn about Safety and efficacy of preoperative adjuvant SOX regimen combined with nivolumab versus FLOT Regimen with nivolumab in HER2-negative Gastric or Gastroesophageal Junction Adenocarcinoma. The main question it aims to answer are:

* Safety and efficacy of preoperative adjuvant SOX regimen combined with nivolumab versus FLOT regimen with nivolumab for the treatment of HER2-negative Gastric or Gastroesophageal Junction Adenocarcinoma.
* Disease-free survival of preoperative adjuvant SOX plus nivolumab and FLOT plus nivolumab for HER2-negative Gastric or Gastroesophageal Junction Adenocarcinoma.

Participants will be divided into two groups to use a FLOT chemotherapy regimen plus nivolumab (one group) and a SOX chemotherapy regimen plus nivolumab (another group). Researchers would compare tumor regression grade, adverse effects and survival benefit of two neoadjuvant regimens.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histopathological confirmation of GC or GEJC.
* 2. Absence of prior anti-tumor treatments, encompassing surgical resection, chemotherapy, radiotherapy, or immunotherapy.
* 3. Age within the range of 18 to 75 years.
* 4. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0-1.
* 5. Absence of concurrent malignancies.
* 6. For patients with resectable GC, those with locally advanced stage III and IVA were clearly included according to the 8th edition of the American Joint Committee on Cancer (AJCC) staging system, and there were no unresectable factors.
* 7. Patients with HER-2 negative.
* 8. Basal information such as hematology and pathological histology was complete.

Exclusion Criteria:

* 1. Refusal of surgical resection subsequent to neoadjuvant therapy.
* 2. Receipt of other ICIs during the study period.
* 3. Receipt of corticosteroids during the study period.
* 4. Have received any anti-tumor therapy such as chemotherapy, radiotherapy, immunotherapy, etc., or have been more than 180 days since the last treatment.
* 5. Confirmed recurrence of GC.
* 6. Hypersensitivity to the study medication.
* 7. Systemic medical conditions contraindicating chemotherapy.
* 8. Psychiatric illnesses contraindicating chemotherapy.
* 9. Acute infections necessitating antibiotic therapy.
* 10. Uncontrolled diabetes mellitus.
* 11. Metastatic disease.
* 12. Severe malnutrition.
* 13. Active autoimmune disorders.
* 14. Pregnancy or lactation.
* 15. Positive serological test for hepatitis B or C virus infection,
* 16. Untreated central nervous system metastases peripheral neuropathy.
* 17. Severe myelosuppression.
* 18. Severe hepatic or renal insufficiency (Child-Pugh C, estimated glomerular filtration rate [eGFR] <30 mL/min).
* 19. Significant cardiac history.
* 20. Patients with a history of allogeneic organ transplantation.
* 21. History of malignancy within the past 5 years (with the exception of curative, localized cancer).
* 22. Patients with multiple factors affecting oral medication.
* 23. Vaccination within 4 weeks prior to the first dose of study drug.
* 24. Patients who have received immune checkpoint inhibitors and develop serious adverse reactions after treatment and need to be permanently disabled.
* 25. The investigator believes that the subject has other serious systemic diseases or other reasons and is not suitable for this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients came from several tertiary hospitals in Xi'an city, Shaanxi Province, and were diagnosed with locally advanced gastric cancer, and the patients would accept either the neoadjuvant SOX+nivolumab or FLOT+nivolumab regimen.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
adverse event | From the preoperative chemotherapy until the occurrence of adverse events, assessed up to 180 days
  adverse event caused by FLOT, SOX or nivolumab treatment, which were coded using the Medical Dictionary Regulatory Activities version 20.1 and adverse event grade according to the National Cancer Institute Common Terminology Criteria for Adverse Events

SECONDARY OUTCOMES:
tumor regression grade | From the surgery to evaluation of tumor regression grade, assessed up to 1 week
  Residual tumor components in post-radiotherapy samples and the proportion of fibrosis
disease-free survival | From date of diagnosis until the first documented recurrence or death, assessed up to 120 months
  from diagnosis to recurrence or death
objective response rate | From the surgery to evaluation of objective response rate, assessed up to 1 week
  objective response rate defined as the proportion of patients with a complete response or partial response to treatment according to Response Evaluation Criteria in Solid Tumors (RECIST).
Duration of response | From the first assessment of the tumor as CR or PR to the first assessment of PD (Progressive Disease) or death from any cause, assessed up to 120 months.
  Duration of response

CONTACTS AND LOCATIONS:
Overall Officials: Jipeng Li, Doctor, Principal Investigator — Xijing Hospital
Locations (3):
- China (3):
  - Tangdu hospital, Xi'an, Shaanxi
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi
  - Xijing hospital, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: No